CLINICAL TRIAL: NCT04191070
Title: A Three Dimensional Comparative Evaluation of Distal Movement of Entire Maxillary Dentition Using Infrazygomatic Crest Miniscrews and Zygomatic Miniplates: A Randomized Clinical Trial
Brief Title: Distalization Using Infrazygomatic Crest Miniscrews and Zygomatic Miniplates: A Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sonal anu
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Class II correction using infrazygomatic crest miniscrews (Experimental): class II correction by distalization using infrazygomatic crest miniscrews (G1)
  Interventions: Device: infrazygomatic miniscrew
- Class II correction using zygomatic miniplates (Experimental): class II correction by distalization using zygomatic miniplates (G2)
  Interventions: Device: zygomatic miniplate

INTERVENTIONS:
Device: infrazygomatic miniscrew — class II correction by distalization using infrazygomatic crest miniscrew
  Arms: Class II correction using infrazygomatic crest miniscrews
Device: zygomatic miniplate — class II correction by distalization using zygomatic miniplate
  Arms: Class II correction using zygomatic miniplates

SUMMARY:
The main objective of this study is to quantify the distal movement of maxillary central incisors and molars achieved with infrazygomatic miniscrews in comparison with zygomatic miniplate anchorage.

DETAILED DESCRIPTION:
Premolar extraction treatment with multibracketed system and reinforced anchorage has been a common modality for correcting maxillary incisor crowding or class II malocclusion due to maxillary protrusion in nongrowing patients. Treatment of class II malocclusion without extraction frequently requires distalization of maxillary molars into class I relation by means of extraoral or intraoral forces.

Extra oral headgear traction is the oldest and most commonly used method to correct class II buccal segment relationship by restricting the forward growth of maxilla and /or distalizing the maxillary molars. This distalizes not only 1st molar but also maxillary 1st and 2nd premolars via transseptal fibers. Headgear is seldom an option in adults due to aesthetics and compliance concerns. The disadvantages of extra-oral appliances have motivated many investigators to develop the mechanics of intraoral molar distalization.

Various intraoral non-compliance appliances like magnets, distal jet, jones jig, pendulum appliance etc. have been used to distalize the maxillary molars. However, in these appliances, anchorage loss characterized by protrusion of maxillary incisors and an increase in overjet is seen. Also, considerable amount of relapse occured when the distalized molars were used as anchorage for the retraction of anteriors and premolar teeth.

Absolute skeletal anchorage available 24 hours a day is an alternative method for molar distalization. It provides stationary anchorage for various tooth movements without the need for active patient compliance and with no undesirable side effects. Inter radicular miniscrews placed between the roots limit the amount of distalization possible as they come in contact with surrounding roots during tooth movement. Also, proximity of miniscrews to the roots may lead to failure of screw anchorage.

Infrazygomatic crest is a site for miniscrew placement. It has been used successfully to provide skeletal anchorage for en-masse anterior retraction, canine retraction, and intrusion of maxillary posterior teeth. Anatomically, it is a pillar of cortical bone at the zygomatic process of maxilla. It has two cortical plates - sinus floor and buccal cortical plate. This allows for bicortical fixation and contributes to better primary stability of miniscrew. A thicker bone allows greater miniscrew biting depth and more osseous contact . A new method for maxillary dentition distalization with miniscrews implanted in the infrazygomatic crest (IZC) region was proposed by Lin. There is no interference with tooth movement by miniscrews placed here and the technique is easy to master .

Miniplates are also fixed at a distance from the root apices, and therefore do not interfere in tooth movement. Their placement and removal however requires a more invasive surgical procedure than those of miniscrews. Until now, there have been only few clinical studies involving group distalization of posterior teeth. Thus little information is available regarding the type of tooth movement that occurs, its limitations and post treatment stability.

Sugawara et al reported that the maxillary 1st molars were moved to the distal by approximately 4mm at crown level by miniplate anchorage. However inconsistent sampling comprising of class I, class II and class III malocclusion failed to throw light on the clinical applicability and treatment planning. Also in this study 2nd molars were extracted in some patients while 3rd molars were extracted in others which might have led to different rates of tooth movement. This study was evaluated on lateral cephalogram in wide-open mouth thus studying the tooth movement in two dimensions only.

Wu X et al(11) reported that mesiobuccal cusp of maxillary 1st molar crowns were moved to the distal by approximately 3.15mm and distobuccal cusp by 2.8mm with miniscrews implanted in the infrazygomatic crest (IZC). However, no attempt was made to evaluate the distalization effect on 2nd molar. Though this study was evaluated with 3D reconstruction module from Cone Beam Computed Tomography, this study did not evaluate the root resorption occuring during treatment.

So far, most distalization studies have used 2-dimensional lateral cephalograms. The disadvantages of this approach include confounded images caused by superimposed anatomic structures and a lack of right and left side information. Although cone-beam computed tomography (CBCT) has disadvantages that include higher doses of radiation, higher cost, and limited availability, these limitations are overcome by the huge amount of data that is provided without distortion or superimposition.

No prospective randomized clinical trial has been carried out on distalization of entire maxillary dentition so far. Also, to the best of our knowledge, no study to evaluate distalization of entire maxillary dentition with Infrazygomatic crest miniscrews in comparison with zygomatic miniplates has been conducted till now.

The purpose of this randomized clinical study is to make a detailed comparison of distalization of entire maxillary dentition using miniscrews implanted in infrazygomatic crest with those of zygomatic miniplates in non-growing patients using Cone Beam Computed Tomography.

MATERIALS AND METHOD Ours is a prospective, non-pharmacological, single blind, randomized clinical study to make a detailed comparison of distalization of entire maxillary dentition using miniscrews implanted in infrazygomatic crest with those of zygomatic miniplates in non-growing patients using Cone Beam Computed Tomography. The present study will be conducted in the Department of Orthodontics and Dentofacial Orthopaedics, in conjunction with Department of Oral and Maxillofacial Surgery, P.G.I.D.S., Pt. B.D.Sharma University of Health Sciences, Rohtak. The study will be carried out after the institutional approval obtained from the ethical committee.

SOURCE OF DATA The sample size consists of 42 subjects selected from the patients attending the regular Out Patient Department at the Department of Orthodontics and Dentofacial Orthopaedics for orthodontic treatment.

TARGET SAMPLE SIZE A sample size of 17 per group for the present study was calculated to detect a clinical difference of 2.3 mm with a standard deviation of 2.3mm (effect size 1.0) at 80% power and 95% confidence interval. To compensate for 20% dropouts the final sample size was calculated to be 21 per group.

INTERVENTION AND DESIGN OF STUDY. The main intervention in this prospective clinical study is the placement of miniscrews at infrazygomatic crest/ zygomatic miniplates after initial leveling and alignment of maxillary dental arch. The study consists of 2 groups with equal allocation of subjects in each group.Group 1 (G1) :- This group will receive infrazygomatic crest miniscrews bilaterally.Group 2 (G2) :-This group will receive zygomatic miniplates bilaterally. Selection of subjects (patients meeting selection criteria).Treatment with 0.022" MBT preadjusted edgewise appliance. Maxillary arch will be stabilized with the help of 0.019" × 0.025" stainless steel.Randomized allocation to 2 groups-G1, G2. Pretreatment diagnostic records including CBCT will be taken before placement of skeletal anchorage devices (infrazygomatic crest miniscrews/ zygomatic miniplates).Maxillary 3rd molars will be extracted, if present. Insertion of skeletal anchorage devices under LA as per the group allocated. Hooks will be soldered on archwire used for stabilizing dentition.Ni-Ti closed coil spring/e-chain will be used to apply force from the skeletal anchorage device to the hooks on the wire.

Patient recalled at 4 weeks interval.Regular follow up of the patient will be done and records including CBCT will be taken on achievement of class I molar relation bilaterally.

CBCT SPECIFICATIONS:During CBCT scan, patients will be instructed to maintain an upright posture and bite on a CT guide plate so as to open the contact between maxillary and mandibular dentition and stabilize the patient. The CBCT scans will be performed using CS 9300 CBCT machine at 85 kV, 4mA current, exposure time of 6.30 seconds, 17 x 6 FOV and voxel size of 180 micro millimeter. All the scans will be performed by the same researcher.Another Cone Beam Computed Tomography will be taken 2 years post retention.

DATA COLLECTION AND CONE BEAM COMPUTED TOMOGRAPHY ANALYSIS The investigator will record the patients' name, address, contact number and other relevant case history records will be taken. Cephalometric radiographs and Cone Beam Computed Tomography and will be recorded before placement of zygomatic miniplates,on achievement of Class I molar relation bilaterally and 2 years post retention for assessment of distalization. These records will be analyzed. The relevant values will be entered in a predesigned format. Soft tissue profile changes between pretreatment and post treatment will be assessed on lateral cephalogram and the raters- orthodontist, laypersons,patients,parents and general dentists will assess changes in facial appearance on a visual analog scale with profile photographs and comparison will be done between the two groups. Patient perception will be assessed using questionare rating by patient regarding various parameters at 1week, 2 weeks, 1 month and 6 months after the placement of zygomatic miniplate or IZC miniscrew. Quality of life will also be assessed using questionnaire rating by patient at pre-treatment, mid-treatment and post treatment. Occlusal status changes between pre and post treatment will be assessed using PAR index(peer assessment rating between 2 groups).

INFORMED CONSENT OF THE PATIENT A valid, informed written consent of the patient or parent/ guardian will be obtained from the patient before registering the patient in this clinical study . Patient will be informed about all the theoretical risks and benefits of the intervention under test .Risks and hazards of radiation during CBCT will also be explained to the patient. The patient will be given 72 hours to discuss the study with his/her family and take the decision regarding participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Non growing patients
* Bilateral Class II molar relationship, defined by at least end-to-end molar relationship.
* No or minor crowding in the mandible.
* Treatment completion without any permanent teeth extracted (excluding third molars).
* Both 1st and 2nd maxillary molars present on the side with a Class II relationship.
* Horizontal to average growth pattern.

Exclusion Criteria:

* Subjects with a history of fixed orthodontic treatment.
* Crossbite
* Vertical growth pattern
* Any systemic disease affecting bone and general growth
* Poor oral hygiene
* Cleft patients
* Patients who fail to follow up or undergo complete treatment

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
distal movement of maxillary molars and central incisors measured in mm at crown and root levels | 28 months
  . distal movement of maxillary molars and central incisors measured in mm at crown and root levels achieved with infrazygomatic crest miniscrew in comparison with zygomatic miniplates on Cone Beam Computed Tomography
root resorption of maxillary teeth | 28 months
  root resorption of maxillary incisors, canines, premolars and molars evaluated on Cone Beam Computed Tomography before and after distalization with infrazygomatic crest miniscrew in comparison with zygomatic miniplates
patient experiences and quality of life with zygomatic miniplates and infrazygomatic crest miniscrews | 34 months
  patient experiences and quality of life with zygomatic miniplates and infrazygomatic crest miniscrew assessed using questionnaires given to patients for evaluating patient attitude,pain perception and quality of life at different time intervals.
soft tissue profile changes | 34 months
  soft tissue profile changes after distalization evaluated on lateral cephalogram and the raters- orthodontist, laypersons,patients,parents and general dentists will assess changes in facial appearance on a visual analog scale with profile photographs
occlusal status comparison | 34 months
  occlusal status changes pre and post treatment will be assessed using PAR index(peer assessment rating between 2 groups)

SECONDARY OUTCOMES:
mandibular plane angle | 28 months
  changes in mandibular plane angle after distalization with infrazygomatic crest miniscrew in comparison with zygomatic miniplates
movement of maxillary central incisors and molars in vertical plane | 28 months
  movement of maxillary central incisors and molars in vertical plane assessed by measuring the perpendicular distance between the incisal edge/ mesio-buccal cusp to the palatal plane on Cone Beam Computed Tomography after distalization with infrazygomatic crest miniscrew in comparison with zygomatic miniplates
transverse changes | 28 months
  intercanine and intermolar changes in transverse plane pre and post distalization will be measured on CBCT
airway changes | 28 months
  Changes in the upper-airway size will be measured by using lateral cephalometric radiographs taken before and after distalization

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol